CLINICAL TRIAL: NCT03004625
Title: Treatment Efficacy and Safety of 12 Weeks of Daclatasvir, Asunaprevir Plus Ribavirin for HCV Genotype 1b Without Baseline NS5A Resistance-associated Variants (DARING)
Brief Title: Daclatasvir, Asunaprevir Plus Ribavirin for HCV Genotype 1b Without NS5A RAV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI444-406
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Arm (Experimental): HCV-1b patients without baseline NS5A resistance-associated variants receiving Daclatasvir (60mg/day) and asunaprevir (100 mg twice daily) plus weight-based ribavirin (1000-1200 mg/d) for 12 weeks. (daclatasvir, asunaprevir plus ribavirin)
  Interventions: Drug: daclatasvir; Drug: asunaprevir; Drug: Ribavirin

INTERVENTIONS:
Drug: daclatasvir — to evaluate the treatment efficacy and safety of the drug in HCV patients
  Other Names: Daklinza
Drug: asunaprevir — to evaluate the treatment efficacy and safety of the drug in HCV patients
  Other Names: Sunvepra
Drug: Ribavirin — to evaluate the treatment efficacy and safety of the drug in HCV patients
  Other Names: Robatrol

SUMMARY:
A single-arm, multi-center study of HCV-1b patients without baseline non-structure protein (NS5A) resistance-associated variants. Daclatasvir (60mg/day) and asunaprevir (100 mg twice daily) plus weight-based ribavirin (1000-1200 mg/d) for 12 weeks will be prescribed.

DETAILED DESCRIPTION:
Twenty-four weeks of Daclatasvir plus Asunaprevir provided a high treatment efficacy in hepatitis C virus genotype 1b (HCV-1b) patients. Patients with non-structural protein 5A (NS5A) resistance associated variants (RAVs) would have an inferior response. The investigators anticipate that12 weeks of daclatasvir and asunaprevir plus ribavirin is highly effective for HCV Genotype 1b patients without baseline NS5A RAVs.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naïve, interferon-experienced, interferon-intolerant or interferon-ineligible, HCV genotype 1b patients with compensated liver disease.
2. Patients with compensated liver cirrhosis will be capped at 40%.

   Cirrhosis is defined as any one of the following:
   * Liver biopsy showing cirrhosis
   * Fibroscan indicative of cirrhosis as evidenced by a result > 12.5 kilopascal

   Absence of cirrhosis is defined as any one of the following:
   * Liver biopsy within 2 years of Screening showing absence of cirrhosis
   * Fibroscan within 6 months of Baseline with a result of ≤ 12.5 kilopascal
3. History of chronic HCV infection > 6 months
4. Aged at least 20 years
5. HCV RNA of 10,000 IU/mL or greater
6. Negative serum or urine pregnancy test result (sensitivity of 25 international units or better) for women with childbearing potential within the 24-hour period before the first dose of study drugs
7. Female patients with childbearing potential must agree to use two reliable forms of effective non-hormonal contraception (i.e., condoms, cervical barriers, intrauterine device, spermicides, or sponge), at least 1 of which must be a physical barrier method, during treatment and for at least 6 months following the last dose of ribavirin.
8. A hormonal contraception (in lieu of non-hormonal) plus a physical barrier method can be used after end of treatment. All men with female partners of childbearing potential must use two reliable forms of effective contraception (combined) during treatment and for 6 months following the last dose of ribavirin
9. Ability to participate and willingness to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

1. The existence of baseline NS5A RAV "Lycine 31 (L31F/I/M)" or "Tyrosine93 (Y93H)", by using direct-sequencing with RAV of > 20%.
2. Hepatitis B virus or HIV co-infection.
3. Patients with experience of ascites, oesophageal varices, or other evidence of hepatic decompensation, and/or hepatocellular carcinoma.
4. History of organ transplantation, except cornea transplantation.
5. Hemoglobin concentration < 12 g/dl for male, 11 g/dl for female
6. Platelet count < 50,000/mm3
7. Prior direct antiviral agents (DAAs) experienced.
8. History of active malignancy within the last 5 years, with the exception of localized or in situ carcinoma (e.g., basal or squamous cell carcinoma of the skin)
9. History of severe cardiac disease (e.g., New York Heart Association Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmia's requiring ongoing treatment, unstable angina or other unstable, uncontrolled or significant cardiovascular disease within 6 months).
10. Poorly controlled diabetes (Hemoglobin A1c value ≥ 8.5%) and endocrine condition.
11. Total bilirubin >2 mg/dL, unless subject has a documented history of Gilbert's disease.
12. Creatinine Clearance (CrCl) <30 mL/min (as estimated by Cockcroft and Gault)
13. Pregnant or lactating women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-11; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
To determine the treatment efficacy (SVR12) of 12 weeks of daclatasvir and asunaprevir plus ribavirin for HCV-1b patients without baseline RAVs | 6 months (including 3 months of treatment and 3 months of post-treatment follow-up peroid
  SVR12 is defined as undetectable HCV RNA 12 weeks throughout 12 weeks of post-treatment follow-up peroid

SECONDARY OUTCOMES:
To evaluate the number of participants with treatment-related adverse events of 12 weeks of daclatasvir and asunaprevir plus ribavirin for HCV-1b patients without baseline RAVs. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, MD., PhD., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical Universsity, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No